CLINICAL TRIAL: NCT05574322
Title: Efficacy of a Foot Strengthening Protocol on Sport Performance Kinetics
Acronym: PRP-Pied-PERF
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: inclusion rate too low
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 21CH247; ANSM (Other: 2022-A00376-37)
Record Dates: First submitted 2022-10-03; First posted 2022-10-10 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Healthy Athletes; Healthy Volonteers
Keywords: Foot strength; resistance training; kinetics,; sprinting; cutting; jumping; sport performance
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: This is a single-center randomized controlled trial (RCT) in 2 parallel groups of athletic participants (18-40 years) in good general health: one receiving an 8-week muscle strengthening program (PRP group), the other not (control group) strengthening program (PRP group), the other not (control group).
Who Masked: Participant
Masking Description: The RCT is divided into 3 distinct periods (see study diagram in Appendix 1): a 4-week control period, an 8-week intervention period and a 4-week follow-up period. This 3-period experimental design was designed to was designed to reduce various methodological biases
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Training group (PRP) (Experimental): Participants benefiting from an 8-week muscle strengthening program (PRP)
  Interventions: Other: Progressive foot strengthening protocol
- Control group (Sham Comparator): Participants in the control group will be asked to maintain their habits and lifestyle (without training program) for the duration of the study.
  Interventions: Other: Control group

INTERVENTIONS:
Other: Progressive foot strengthening protocol — This interventional group will perform the foot strengthening protocol (PRP) with physical tests as :
  * Maximum muscle strength of the foot
  * Foot muscle morphology
  Arms: Training group (PRP)
Other: Control group — The control group will not perform the foot strengthening protocol and will continue with all their daily activities with no change in lifestyle.
  Arms: Control group

SUMMARY:
This randomized controlled trial aims to explore the effect of a foot strengthening protocol on toe flexion strength, foot deformation and morphology as well as kinetics during sprinting, cutting and jumping in healthy athletes (18-40 completed years). The study consists of a 4 weeks control period, followed by 8 weeks intervention period and 4 weeks follow up

DETAILED DESCRIPTION:
During the first period participants are unaware of their allocation, while in the intervention period they will be allocated to a train intervention or a control group (habits maintenance). The primary outcome is the toes maximal voluntary isometric plantarflexion. The treatment effectiveness estimand is the same as in a pretest-posttest case control study, considering the end of the control period as pre-point. An estimation of the individual variability in response to the treatment will be provided.

ELIGIBILITY:
Inclusion criteria :

* To be affiliated in the federation of one of the following sports : soccer, handball, rugby, basketball or track and field;
* To practice their respective sport more than two times per week;
* Be affiliated or beneficiary of a social security insurance;
* Having freely given their written consent after having been informed of the purpose, the procedure and the potential risks involved.
* Licensed in a tennis club (FFT) and in a volleyball club (FFVolley)

Exclusion criteria :

* Use of pharmacological therapy to match gander identity;
* Have an abnormal range of motion of the toes and/or ankle;
* Have any kind of ankle or foot pain (self-defined and self-reported by the FAAM questionnaire) in the previous 6 months;
* Have a previous injury or surgery of the lower limb in the previous 6 months;
* Have a neurological or vestibular deficit that may affect walking or balance (lumbar-sacral radiculopathy, peripheral nerve pathology, Marfan or Eehlers-Danlos syndrome, etc.);
* Have contraindication to neuromuscular electrical stimulation (pacemaker, seizure disorders, pregnancy);
* Have a previous foot strengthening experience in the past 6 months for at least 2 weeks and more than one session per week;
* Participate at the same time in another medical interventional experiment or have participated in such a study in the 30 days preceding this study;
* Being unable to understand the purpose and conditions of the study, and to give consent;
* Being deprived of liberty or under guardianship.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2023-02-03 (Actual); Primary Completion 2024-02-14 (Actual); Study Completion 2024-06-13 (Actual)

PRIMARY OUTCOMES:
maximal isometric joint flexion muscle strength MTP (in N) | Change from baseline to Week 18
  It will be measured using an ergometer composed of a 3-dimensional force sensor (Nano 25, ATI Industrial Automation, Garner, NC) during the 3 periods of the randomized controlled trial (control, intervention and follow-up) and repeatedly each week during the intervention protocol.

SECONDARY OUTCOMES:
Foot deformity | Change from baseline to Week 18
  It's a composite outcome :
  Foot deformity will be assessed with the help of the system (Arch Height Index Measurement System, JAKTOOL Corporation, Cranberry, NJ) measuring the following variables (in cm): height of the navicular, total length of the foot, truncated length of the foot, width of the medial foot and height of the dorsal arch when the participant is sitting and then when standing on one foot.
Foot posture | Change from baseline to Week 18
  Foot posture will be measured using the Foot Posture Index (FPI-6).
Morphology of the foot muscles | Change from baseline to Week 18
  The morphology of the foot muscles will be evaluated by measuring with the AixPlorer Ultrasonic scanner, version 6.1.1; Supersonic Imagine, Aix-en-Provence, France.
general stiffness of the foot-ankle complex | Change from baseline to Week 18
  The general stiffness of the foot-ankle complex will be evaluated using an optical measurement system (Optojump Next, Microgate, Bolzano, 113 Italy) during 6 maximal jumps with knees stretched.
propulsion impulse during sprinting | Change from baseline to Week 18
  The propulsion impulse during sprinting will be evaluated using 6 force platforms embedded in the ground (Kistler, Winterhur, Switzerland) allowing to collect kinetic parameters of forces in the 3 dimensions of space at a sampling frequency of 2000 Hz.
propulsion impulse during jumps | Change from baseline to Week 18
  The propulsion impulse during jumps will be evaluated using 2 force platforms embedded in the ground under each foot (Kistler, Winterhur, Switzerland) to collect kinetic force parameters in all 3 spatial dimensions during vertical and horizontal jumps at a sampling frequency of 2000 Hz.
propulsion impulse during direction changes | Change from baseline to Week 18
  The propulsion impulse during direction changes will be evaluated using a ground embedded force platform (Kistler, Winterhur, Switzerland) to collect force kinetic parameters in all 3 spatial dimensions during 90° direction changes at a sampling rate of 2000 Hz.

CONTACTS AND LOCATIONS:
Overall Officials: Pascal EDOUARD, PhD, Principal Investigator — Centre Hospitalier Universitaire de Saint Etienne
Locations (1):
- CHU de Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No